CLINICAL TRIAL: NCT00042536
Title: Effects of Alpha-2 Adrenergic and Opiate Receptor Blockade on Sexual Function in Healthy Male Volunteers
Brief Title: Effects of Yohimbine and Naltrexone on Sexual Function
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 020262; 02-M-0262
Record Dates: First submitted 2002-07-31; First posted 2002-08-01 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2004-04

CONDITIONS: Erectile Dysfunction
Keywords: Yohimbine; Naltrexone; Sexual Function; Erectile Dysfunction; Alpha-2 Adrenoreceptor; Opiate Receptor; Male Impotence; ED; Healthy Volunteer; HV; Normal Control
MeSH Terms: conditions — Erectile Dysfunction | interventions — Naltrexone; Yohimbine

INTERVENTIONS:
Drug: Naltrexone HCL/ Yohimbine HCL

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of the drugs yohimbine and naltrexone in treating men with erectile dysfunction (ED) (the inability to achieve or maintain penile erection for satisfactory sexual performance).

ED is a medical and psychological problem that is usually associated with increased age. Evidence suggests that specific neurotransmitter systems are involved in the regulation of sexual function. Yohimbine and naltrexone are drugs that may influence these neurotransmitter systems. This study will use different doses of yohimbine and fixed doses of naltrexone to determine their effectiveness in treating ED.

Participants in this study will be screened with a medical history, physical examination, blood and urine tests, and an electrocardiogram (ECG). The study will consist of three outpatient visists.

DETAILED DESCRIPTION:
Erectile dysfunction (ED) is a relevant medical and psychological problem for males, and is usually associated with increased age. There is substantial evidence available suggesting that noadrenergic and opiate transmitter systems are involved in regulation of sexual function. The objective of the present study is to evaluate the effects and safety of a potential novel treatment combination for ED consisting of both, the alpha-adrenoreceptor antagonist yohimbine, and the opiate antagonist naltrexone. The study uses a three-phase, double-blind, placebo-controlled cross-over design. Healthy, male volunteers will participate. The effects of differing dosages of yohimbine (10 mg versus 20 mg) and a fixed dose of naltrexone (50 mg) on penile tumescene and rigidity, and sexual arousal are assessed in a placebo-controlled design. The anticipated risks of the study are considered minimal in relation to the importance of our increased knowledge about regulation of physiological and psychological aspects of regulation of sexual function and dysfunction. This novel treatment combination could be later also applied to patients with ED of different origin, e.g. organic, psychogenic, and mixed causes.

ELIGIBILITY:
INCLUSION CRITERIA

Subjects must be medically healthy and free of mental illness, take no medication, and must report no problems with their sexual function. They are required to be sexually active, including successful penetrative sexual intercourse acts.

For assessments of sexual function before and after the study subjects are required to complete a detailed daily diary recording their erectile activity for 7 days before the first study session, and for 7 days after completion of the study.

EXCLUSION CRITERIA

Persons having taken antidepressant or other medications likely to alter monoamine neurochemistry or cerebrovascular and cardiovascular function within 6 months prior to the study will be excluded.

Individuals will also be excluded if they have: a) evidence for an axis I psychiatric disorder (DSM-IV criteria), b) medical or neurological illnesses likely to affect physiology or anatomy, c) a history of drug (including BZDs) or alcohol abuse within 1 year or a lifetime history of alcohol or drug dependence (DSM IV criteria), d) smokers, e) diagnosis of a sexual disorder, f) criminal history.

Persons must exhibit no or only moderate alcohol use. Persons with current or previous regular use ( more than 4 weeks) of BZDs and excessive use of alcohol (more than 8 ounces/day) in the past or presence are ineligible to participate, as such drug use confound the results.

Individuals beyond age 50 are excluded because subjects beyond age 50 have a far greater likelihood of showing subtile, albeit clinical irrelevant disturbances in erectile function.

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40
Dates: Start 2002-07; Study Completion 2004-04

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Mental Health (NIMH), Bethesda, Maryland, United States

REFERENCES:
- [Background] NIH Consensus Conference. Impotence. NIH Consensus Development Panel on Impotence. JAMA. 1993 Jul 7;270(1):83-90. No abstract available. PMID 8510302
- [Background] Feldman HA, Goldstein I, Hatzichristou DG, Krane RJ, McKinlay JB. Impotence and its medical and psychosocial correlates: results of the Massachusetts Male Aging Study. J Urol. 1994 Jan;151(1):54-61. doi: 10.1016/s0022-5347(17)34871-1. PMID 8254833
- [Background] Blanker MH, Bosch JL, Groeneveld FP, Bohnen AM, Prins A, Thomas S, Hop WC. Erectile and ejaculatory dysfunction in a community-based sample of men 50 to 78 years old: prevalence, concern, and relation to sexual activity. Urology. 2001 Apr;57(4):763-8. doi: 10.1016/s0090-4295(00)01091-8. PMID 11306400